## **INFORMED CONSENT FORM – MOVE CLINICAL STUDY**

Protocol ID: MOVE-001/2025 | Version 1.0 | Date: June 15,

2024

Study Title: Movement-Oriented Velocity of Engagement

(MOVE) Protocol

**Authority** 

Principal Investigator: Dr. Neeraj Mehta, Ph.D. | MMSx

Ethics Approval: Institutional Research Ethics Board (IREB

Approval No: IREB/2024/067)

Organization: MMSx Authority – Institute for Movement

Mechanics & Biomechanics Research

Address: 940 Vauxhill Lane, Powell, Ohio 43065, USA

Contact: info@mmsxauthority.com

**MMSx Authority — IREB** 

IREB Home **MOVE Dashboard** 

### **Participant Informed Consent Form**

#### **Study Title & Sponsor**

#### M.O.V.E. Protocol — Movement-Oriented Velocity of Engagement

Sponsor: MMSx Authority (with BodyGNTX USA, GFFI India, IIKBS Affiliate; academic collaboration with ASFU)

#### **Purpose of the Study**

To evaluate the safety and effectiveness of an early-mobilization rehabilitation approach (MOVE) for musculoskeletal pain and recovery.

#### **Procedures**

- Assessment at baseline, week-2, week-4, and week-8 (pain, function, balance, activity tolerance).
- Participation in MOVE sessions: Mobilize, Optimize Load, Validate Neural Control, Energize Recovery.
- Home program: brief daily mobility and walking/cycling (20–30 minutes as tolerated).

## **Risks & Discomforts**

Temporary soreness or symptom flare may occur. Serious risks are unlikely but include falls or strain. You should report any symptoms to your investigator immediately.

#### **Benefits** Potential reduction in pain, improved function, and faster return to activities.

Benefits are not guaranteed.

## Usual care, rest/medication, or other rehabilitation options. You may discuss

**Alternatives** 

alternatives with your clinician.

## Your data will be de-identified for analysis. Records may be reviewed by the

Confidentiality

MMSx IREB for monitoring.

## benefits.

**Voluntary Participation & Withdrawal** 

Participation is voluntary. You may withdraw at any time without penalty or loss of

# No direct payment is offered. There are no costs beyond your usual travel/time.

**Compensation & Costs** 

**Contacts for Questions** 

Study team: info@mmsxauthority.com. For rights as a participant, contact MMSx

# IREB.

**Consent & Authorization** 

Participant Signature / Date Witness Signature / Date

Investigator / Authorized Designee Signature / Date

By signing, I confirm I have read and understood this consent form and agree to participate.

**Download PDF**